CLINICAL TRIAL: NCT05440149
Title: The Postoperative Radiotherapy After Breast Conserving Surgery or Mastectomy in N1 Breast Cancer Patients: a Prospective, Multicenter, Phase III Clinical Trial
Brief Title: The Postoperative Radiotherapy in N1 Breast Cancer Patients
Acronym: PORT-N1
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Kyung Hwan Shin, Professor, Chairman, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0720222005
Record Dates: First submitted 2022-06-27; First posted 2022-06-30 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Radiotherapy; Breast Cancer
Keywords: Breast Cancer; Radiotherapy; Omission; Breast Conserving Surgery; Mastectomy; TNM pathologic stage N1
MeSH Terms: conditions — Breast Neoplasms | interventions — Mastectomy; Mastectomy, Segmental

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The Control group (Active Comparator): * If patients received mastectomy, post-mastectomy radiation therapy (PMRT) should be performed.
  * If patients received breast conserving surgery (BCS), whole breast irradiation (WBI) + Regional radiotherapy (RT) should be performed.
  Interventions: Radiation: PMRT for mastectomy / WBI + Regional RT for BCS
- The Experimental group (Experimental): * If patients received mastectomy, No PMRT should be performed.
  * If patients received BCS, WBI alone should be performed.
  Interventions: Radiation: No PMRT for mastectomy / No regional RT for BCS

INTERVENTIONS:
Radiation: No PMRT for mastectomy / No regional RT for BCS — * Regional RT includes high-tangent field, and can include undissected axilla.
  * The definition of high-tangent is that the upper margin of the radiotherapy field located within 2 cm of the humeral head to include axillary levels I and II.
  * Both hypofractionated and conventionally fractionated radiation therapy are allowed, and 3-dimensional or intensity modulated radiotherapy are allowed. The electron beam can also be used.
  Arms: The Experimental group
Radiation: PMRT for mastectomy / WBI + Regional RT for BCS — * Regional RT includes high-tangent field, and can include undissected axilla.
  * The definition of high-tangent is that the upper margin of the radiotherapy field located within 2 cm of the humeral head to include axillary levels I and II.
  * Both hypofractionated and conventionally fractionated radiation therapy are allowed, and 3-dimensional or intensity modulated radiotherapy are allowed. The electron beam can also be used.
  Arms: The Control group

SUMMARY:
This study is a multicenter, randomized, phase 3 clinical trial in patients with breast cancer, randomizing radiotherapy group (postmastectomy radiation therapy (PMRT)/whole breast irradiation plus regional radiotherapy (WBI+regional RT) versus and no PMRT/WBI alone group. This is a non-inferiority study aiming that there is no significant difference in the 7-year disease-free survival rate between the two groups.

DETAILED DESCRIPTION:
1:1 randomization to the control group and experimental group, stratified by the type of surgery (breast-conserving surgery (BCS) versus mastectomy) and the type of histologic type (triple negative breast cancer (TNBC) versus non-TNBC)

The control group:

* If patients received BCS, WBI+Regional RT
* If patients received mastectomy, PMRT

The experimental group:

* If patients received breast conserving surgery, WBI alone
* If patients received mastectomy, No PMRT

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 19 years or older.
* A female patient who underwent breast-conserving surgery or mastectomy for invasive breast cancer.
* Patient with stage pN1 after surgery on histopathologic examination.

  * However, if mastectomy was performed, 5 or more nodes should be resected in the case of 1 positive node, and axillary lymph node dissection (ALND) should be performed in case of 2 or 3 positive nodes.
* Patients undergoing or planning to undergo hormone therapy in the case of hormone receptor positive.
* Patients who have received or are expected to undergo targeted therapy in the case of human epidermal growth factor receptor(HER)-2 positive.
* Patients with Eastern Cooperative Oncology Group (ECOG) Scale 0-2.
* Patients who agreed to participate in the study.

Exclusion Criteria:

* Patients who have received prior [neoadjuvant] chemotherapy.
* Patients receiving radiation therapy for salvage or palliative purposes.
* Patients with stage T4.
* Patients with ipsilateral supraclavicular and internal mammary lymph node metastases or distant metastases.
* Male breast cancer patient.
* Patients who have previously received radiation therapy to the ipsilateral breast or supraclavicular region.
* Patients having a history of cancer other than thyroid cancer, cervical carcinoma in situ, or skin cancer.
* Patients diagnosed with ductal breast carcinoma in situ, lobular carcinoma in situ, phyllodes, metaplastic cancer, or benign tumors based on histological diagnosis.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1106 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2033-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease-Free Survival | 7-Year
  Time from randomization to local recurrence, regional recurrence, distant metastases, or breast cancer-related death.

SECONDARY OUTCOMES:
Locoregional-Recurrence Free Survival | 7-Year
  Time from randomization to recurrence of tumors in the ipsilateral chest wall, breast or regional lymph nodes (ipsilateral axillary/internal mammary/supraclavicular lymph nodes) or breast cancer-related death.
  ** Recurrence should be confirmed by histological diagnosis, but local recurrence can be diagnosed by clinical examination only when regional/remote or distant metastases already exist.
Distant Metastases Free Survival | 7-Year
  Time from randomization to the development of distant metastases or breast cancer-related death.
Overall Survival | 7-Year
  Time from randomization to the death due to any cause.

OTHER OUTCOMES:
Dermatitis | Every 6 month during 1 years, then every 1 year till 7 years after randomization
  Common Terminology Criteria for Adverse Events (CTCAE) 5.0 Scale
Radiation-related pneumonitis | Every 6 month during 1 years, then every 1 year till 7 years after randomization
  Common Terminology Criteria for Adverse Events (CTCAE) 5.0 Scale
Major complication rate for reconstructed breast | Every 6 month during 1 years, then every 1 year till 7 years after randomization
  For patients who received breast reconstruction after mastectomy
Occurence of contralateral in-situ or invasive breast cancer | Every 6 month during 1 years, then every 1 year till 7 years after randomization
  Pathologic confirmation
Major cardiac event | Every 6 month during 1 years, then every 1 year till 7 years after randomization
  Myocardial infarction / Ischemic heart failure / Unstable angina / Sudden death
Ipsilateral rib fracture | Every 6 month during 1 years, then every 1 year till 7 years after randomization
  Symptom or radiologic diagnosis
Arm Lymphedema | Every 6 month during 1 years, then every 1 year till 7 years after randomization
  Symptom / Diagnosis from the related-department (e.g. rehab) / Expert opinion

CONTACTS AND LOCATIONS:
Overall Officials: Kyung Hwan Shin, MD. PhD., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Jongro-gu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee TH, Chang JH, Jang BS, Kim JS, Kim TH, Park W, Kim YB, Kim SS, Han W, Lee HB, Shin KH. Protocol for the postoperative radiotherapy in N1 breast cancer patients (PORT-N1) trial, a prospective multicenter, randomized, controlled, non-inferiority trial of patients receiving breast-conserving surgery or mastectomy. BMC Cancer. 2022 Nov 16;22(1):1179. doi: 10.1186/s12885-022-10285-0. PMID 36384573